CLINICAL TRIAL: NCT05832853
Title: Hybrid Exercise Program is Frail Elderly Need: Effectiveness on the Physical Abilities and Clinical Assistance From White Box Modeling
Brief Title: A Study of the Intervention Effect of a Hybrid Exercise Program on Frail Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang Yang, Prof. Dr. (Other)
Responsible Party: Sponsor-Investigator, Guang Yang, Prof. Dr., Prof.Dr., Northeast Normal University
Organization: Northeast Normal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CCEE2018
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Frail Elderly Syndrome
Keywords: frailty; exercise intervention
MeSH Terms: conditions — Frailty | interventions — Resistance Training; Endurance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wu Qin Xi exercise (Experimental): The training schedule for Wu Qin Xi consisted of two phases: the first phase lasted for eight weeks, while the second phase lasted for 16 weeks. In the first phase, Wu Qin Xi group was given twice repetitions of the intervention. The second phase consisted of three repetitions of the Wu Qin Xi group.
  Interventions: Behavioral: Wu Qin Xi exercise
- Wu Qin Xi, resistance training and endurance training (Experimental): The trial was divided into three cycles, each lasting eight weeks. Participants performed a hybrid program of Wu Qin Xi exercise, resistance training and endurance training of varying duration and intensity in each cycle. Each session lasted one hour, three times a week for 24 weeks.
  Interventions: Behavioral: Wu Qin Xi, resistance training and endurance training
- Resistance training and endurance training (Experimental): The trial was divided into three cycles, each lasting eight weeks. Participants performed a hybrid program of resistance training and endurance training of varying duration and intensity in each cycle. Each session lasted one hour, three times a week for 24 weeks.
  Interventions: Behavioral: Resistance training and endurance training

INTERVENTIONS:
Behavioral: Wu Qin Xi exercise — The training schedule for Wu Qin Xi consisted of two phases: the first phase lasted for eight weeks, while the second phase lasted for 16 weeks. In the first phase, Wu Qin Xi group was given twice repetitions of the intervention. The second phase consisted of three repetitions of the Wu Qin Xi group. Participants warmed up for 20 min prior to the intervention and cooled down for 10 min at the end.
  Arms: Wu Qin Xi exercise
Behavioral: Wu Qin Xi, resistance training and endurance training — During the first 8 weeks, the training consists of learning and consolidating the movements of the Wu Qin Xi. In the second 16 weeks, participants perform a full set of movement exercises. Each resistance training session contained two lower-body exercises (seated calf raises and hip abduction) and three upper-body exercises (lateral pull downs, biceps curls, and triceps push downs) and two sets for each exercise. Endurance training is performed by continuous walking on an undisturbed indoor track for 15 min. Participants warmed up for 20 min prior to the intervention and cooled down for 10 min at the end.
  Arms: Wu Qin Xi, resistance training and endurance training
Behavioral: Resistance training and endurance training — Each resistance training session contained two lower-body exercises (seated calf raises and hip abduction) and three upper-body exercises (lateral pull downs, biceps curls, and triceps push downs) and three sets for each exercise. Endurance training is performed by continuous walking on an undisturbed indoor track for 30 min. Participants warmed up for 20 min prior to the intervention and cooled down for 10 min at the end.
  Arms: Resistance training and endurance training

SUMMARY:
The declining physical condition of frail elderly is becoming an ugent problem. Although the exercise intensity of Wu Qin Xi appears to be low, it is highly effective in the older individuals. Inspired by the characteristics and functions of Wu Qin Xi, we designed a brand new exercise intervention training program among frail older people, which incorporates Wu Qin Xi, strength exercises and endurance exercises to improve physical fitness, and even reverse the condition of frailty. Furthermore, to improve utility in clinical practice, we innovatively employed machine learning simulations to infer the condition of older adults and predict their level of frailty after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. a Fried frailty phenotype score of 3-5 points;
2. could walk for at least 6 min without support;
3. had not been able to walk in the past year other training.

Exclusion Criteria:

1. people who have a past mental illness or serious psychological issues which make it difficult to obey orders;
2. people who have had neurological disorders within the last six months;
3. people who must regularly participate in other training programs during the study period;
4. people who struggle to walk normally due to significant muscle and skeletal injuries and continuous joint discomfort.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Assessing the endurance of frail older adults using the six-minute walk test | Month 6
  Assessment of endurance in frail older adults before and after intervention using the six-minute walk test
Assessing the speed of frail older adults using the ten-meter maximum walk speed | Month 6
  Assessment of speed in frail older adults before and after intervention using ten-meter maximum walk speed.
Using handgrip strength tests to assess strength in frail older adults. | Month 6
  Using handgrip strength tests to assess strength in frail older adults before and after intervention
Assessment of balance in frail older adults using Time Up and Go Test. | Month 6
  Assessment of balance in frail older adults before and after intervention using Time Up and Go Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Center of Exercise Epidemiology, Changchun, Jilin, China

REFERENCES:
- [Derived] Wei M, He S, Meng D, Yang G, Wang Z. Hybrid Exercise Program Enhances Physical Fitness and Reverses Frailty in Older Adults: Insights and Predictions from Machine Learning. J Nutr Health Aging. 2023;27(10):894-902. doi: 10.1007/s12603-023-1991-0. PMID 37960913